CLINICAL TRIAL: NCT02929329
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of Omecamtiv Mecarbil on Mortality and Morbidity in Subjects With Chronic Heart Failure With Reduced Ejection Fraction (GALACTIC-HF)
Brief Title: Registrational Study With Omecamtiv Mecarbil (AMG 423) to Treat Chronic Heart Failure With Reduced Ejection Fraction
Acronym: GALACTIC-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20110203; 2016-002299-28 (EudraCT Number)
Record Dates: First submitted 2016-09-30; First posted 2016-10-11 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — omecamtiv mecarbil; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omecamtiv Mecarbil (Experimental): Participants received oral omecamtiv mecarbil (OM) twice daily in addition to standard heart failure therapy. The starting dose of OM was 25 mg; At week 4, participants with week 2 OM predose plasma concentrations < 200 ng/mL had their dose increased to 50 mg BID; participants with week 2 predose plasma concentrations ≥ 200 and < 300 ng/mL had their dose increased to 37.5 mg BID and participants with week 2 predose plasma concentrations ≥ 300 ng/mL and < 1000 ng/mL maintained a 25 mg BID dosing regimen.
  Interventions: Drug: Omecamtiv Mecarbil; Drug: Standard of Care
- Placebo (Placebo Comparator): Participants received matching placebo tablets twice a day in addition to standard heart failure therapy.
  Interventions: Drug: Placebo; Drug: Standard of Care

INTERVENTIONS:
Drug: Omecamtiv Mecarbil — Omecamtiv mecarbil tablets for oral administration
  Other Names: AMG 423
  Arms: Omecamtiv Mecarbil
Drug: Placebo — Matching placebo tablets
  Arms: Placebo
Drug: Standard of Care — Participants were required to be optimally managed with standard of care therapies for chronic HF (eg, beta blockers, renin angiotensin aldosterone system inhibitors), consistent with regional clinical practice guidelines, unless contraindicated.

SUMMARY:
The purpose of this study is to determine if treatment with omecamtiv mecarbil when added to standard of care is well tolerated and superior to placebo in reducing the risk of cardiovascular death or heart failure events in adults with chronic heart failure with reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
This study was conducted by Amgen as the IND holder, with Cytokinetics as a collaborator. Due to the termination of the collaboration agreement between Amgen and Cytokinetics in May 2021 and subsequent transfer of the omecamtiv mecarbil IND from Amgen to Cytokinetics, Cytokinetics is now listed as the sponsor.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has provided informed consent
* Male or female, ≥ 18 to ≤ 85 years
* History of chronic heart failure (HF), defined as requiring treatment for HF for a minimum of 30 days before randomization
* Left ventricle ejection fraction (LVEF) ≤ 35%, per subjects most recent medical record, within 12 months prior to screening.
* New York Heart Association (NYHA) class II to IV at most recent screening assessment.
* Managed with HF standard of care (SoC) therapies consistent with regional clinical practice guidelines according to investigator judgment of subject's clinical status
* Current hospitalization with primary reason of HF OR one of the following events within 1 year of screening: hospitalization with primary reason of HF; urgent visit to emergency department (ED) with primary reason of HF.
* Elevated B-type natriuretic peptide (BNP) or n-terminal-prohormone brain natriuretic peptide (NT-proBNP)

Other Inclusion Criteria May apply

Key Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study, or < 30 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Malignancy within 5 years prior to randomization with the following exceptions: localized basal or squamous cell carcinoma of the skin, cervical intraepithelial neoplasia, stage 1 prostate carcinoma, breast ductal carcinoma in situ.
* Subject has known sensitivity to any of the products or components to be administered during testing

Other Exclusion Criteria May apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8256 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (809):
- United States (252):
  - Research Site, Birmingham, Alabama
  - Research Site, Fort Payne, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Scottsboro, Alabama
  - Research Site, Tuscumbia, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Burbank, California
  - Research Site, Carmichael, California
  - Research Site, Fresno, California
  - Research Site, Huntington Beach, California
  - Research Site, Loma Linda, California
  - Research Site, Long Beach, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Redondo Beach, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, San Pedro, California
  - Research Site, Santa Ana, California
  - Research Site, Santa Rosa, California
  - Research Site, Stanford, California
  - Research Site, Stockton, California
  - Research Site, Torrance, California
  - Research Site, Tustin, California
  - Research Site, Ventura, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, West Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Altamonte Springs, Florida
  - Research Site, Aventura, Florida
  - Research Site, Bay Pines, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Crystal River, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Doral, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Naples, Florida
  - Research Site, Ocala, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tampa, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, ‘Aiea, Hawaii
  - Research Site, Arlington Heights, Illinois
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Fairview Heights, Illinois
  - Research Site, Hazel Crest, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Merrillville, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Richmond, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Overland Park, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Crestview Hills, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, West Monroe, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Biddeford, Maine
  - Research Site, Portland, Maine
  - Research Site, Scarborough, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Prince Frederick, Maryland
  - Research Site, Salisbury, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Haverhill, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Grand Blanc, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Midland, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Port Gibson, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Jefferson City, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, North Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Lebanon, New Hampshire
  - Research Site, Eatontown, New Jersey
  - Research Site, Moorestown, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Ridgewood, New Jersey
  - Research Site, Somerset, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Cortlandt Manor, New York
  - Research Site, Johnson City, New York
  - Research Site, Kingston, New York
  - Research Site, Laurelton, New York
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Roslyn, New York
  - Research Site, Saratoga Springs, New York
  - Research Site, Stony Brook, New York
  - Research Site, The Bronx, New York
  - Research Site, Valhalla, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Cary, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Lenoir, North Carolina
  - Research Site, Lumberton, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Tabor City, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Wiloughby, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Abington, Pennsylvania
  - Research Site, Altoona, Pennsylvania
  - Research Site, Butler, Pennsylvania
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Jersey Shore, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Yardley, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Warwick, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Fort Mill, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Germantown, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Oak Ridge, Tennessee
  - Research Site, Powell, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Carrollton, Texas
  - Research Site, Dallas, Texas
  - Research Site, Denison, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Sam Houston, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Galveston, Texas
  - Research Site, Gonzales, Texas
  - Research Site, Houston, Texas
  - Research Site, Huntsville, Texas
  - Research Site, Lubbock, Texas
  - Research Site, McKinney, Texas
  - Research Site, Odessa, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tomball, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Farmington, Utah
  - Research Site, Murray, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Burlington, Vermont
  - Research Site, White River Junction, Vermont
  - Research Site, Charlottesville, Virginia
  - Research Site, Leesburg, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Puyallup, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Huntington, West Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Green Bay, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Manitowoc, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Waukesha, Wisconsin
- Argentina (23):
  - Research Site, Bahía Blanca, Buenos Aires
  - Research Site, CABA, Buenos Aires
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, Coronel Suárez, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Merlo, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Ramos Meija, Buenos Aires
  - Research Site, San Fernando, Buenos Aires
  - Research Site, San Isidro, Buenos Aires
  - Research Site, San Martín, Buenos Aires
  - Research Site, San Nicolás de los Arroyos, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Villa María, Córdoba Province
  - Research Site, Santa Rosa, La Pampa Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Venado Tuerto, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Salta
  - Research Site, Santa Fe
- Australia (17):
  - Research Site, Garran, Australian Capital Territory
  - Research Site, Concord, New South Wales
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Chermside, Queensland
  - Research Site, Herston, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Ashford, South Australia
  - Research Site, Bedford Park, South Australia
  - Research Site, Fullarton, South Australia
  - Research Site, Woodville South, South Australia
  - Research Site, Bundoora, Victoria
  - Research Site, Frankston, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Richmond, Victoria
  - Research Site, Murdoch, Western Australia
- Austria (7):
  - Research Site, Feldkirch
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Sankt Pölten
  - Research Site, Vienna
  - Research Site, Villach
- Belgium (7):
  - Research Site, Aalst
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Lodelinsart
  - Research Site, Roeselare
- Brazil (18):
  - Research Site, Brasília, Federal District
  - Research Site, Goiânia, Goiás
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Uberlândia, Minas Gerais
  - Research Site, Curitiba, Paraná
  - Research Site, Londrina, Paraná
  - Research Site, Natal, Rio Grande do Norte
  - Research Site, Canoas, Rio Grande do Sul
  - Research Site, Passo Fundo, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Aracaju, Sergipe
  - Research Site, Campinas, São Paulo
  - Research Site, Marília, São Paulo
  - Research Site, Ribeirão Preto, São Paulo
  - Research Site, São José do Rio Preto, São Paulo
  - Research Site, São Paulo, São Paulo
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (4):
  - Research Site, Haskovo
  - Research Site, Pleven
  - Research Site, Sandanski
  - Research Site, Sofia
- Canada (26):
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, New Westminster, British Columbia
  - Research Site, North Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, London, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Jean-sur-Richelieu, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Terrebonne, Quebec
- Chile (6):
  - Research Site, Temuco, Cautín
  - Research Site, Talcahuano, Concepción
  - Research Site, Viña del Mar, Región de Valparaíso
  - Research Site, San Miguel, Santiago Metropolitan
  - Research Site, Osorno
  - Research Site, Santiago
- China (30):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Haikou, Hainan
  - Research Site, Harbin, Heilongjiang
  - Research Site, Luoyang, Henan
  - Research Site, Xinxiang, Henan
  - Research Site, Zhengzhou, Henan
  - Research Site, Hengyang, Hunan
  - Research Site, Xiangtan, Hunan
  - Research Site, Hohhot, Inner Mongolia
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Wuxi, Jiangsu
  - Research Site, Xuzhou, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Xi'an, Shaanxi
  - Research Site, Heze, Shandong
  - Research Site, Jinan, Shandong
  - Research Site, Jining, Shandong
  - Research Site, Qingdao, Shandong
  - Research Site, Taiyuan, Shanxi
  - Research Site, Yuncheng, Shanxi
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Ürümqi, Xinjiang
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Linhai, Zhejiang
  - Research Site, Ningbo, Zhejiang
  - Research Site, Beijing
  - Research Site, Shanghai
- Colombia (8):
  - Research Site, Medellín, Antioquia
  - Research Site, Barranquilla, Atlántico
  - Research Site, Manizales, Caldas Department
  - Research Site, Cartagena, Departamento de Bolívar
  - Research Site, Armenia, Quindío Department
  - Research Site, Bucaramanga, Santander Department
  - Research Site, Cali, Valle del Cauca Department
  - Research Site, Bogota D.C.
- Czechia (26):
  - Research Site, Beroun
  - Research Site, Brandýs nad Labem
  - Research Site, Brno
  - Research Site, Frýdek-Místek
  - Research Site, Havlíčkův Brod
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Karlovy Vary
  - Research Site, Kladno
  - Research Site, Klatovy IV
  - Research Site, Kolin III
  - Research Site, Liberec
  - Research Site, Louny
  - Research Site, Mariánské Lázně
  - Research Site, Mohelnice
  - Research Site, Opava
  - Research Site, Ostrava
  - Research Site, Polička
  - Research Site, Prague
  - Research Site, Praha 5 - Smichov
  - Research Site, Pribram VIII
  - Research Site, Svitavy
  - Research Site, Teplice
  - Research Site, Uherské Hradiště
  - Research Site, Zlín
  - Research Site, Znojmo
- Denmark (9):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Esbjerg
  - Research Site, Glostrup Municipality
  - Research Site, Hellerup
  - Research Site, Hillerød
  - Research Site, Køge
  - Research Site, Odense
  - Research Site, Svendborg
- France (24):
  - Research Site, Béziers
  - Research Site, Caen
  - Research Site, Chambray-lès-Tours
  - Research Site, Corbeil-Essonnes
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Grenoble
  - Research Site, Le Chesnay
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Montauban
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Saint-Denis
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Valenciennes
- Germany (21):
  - Research Site, Bad Neuheim
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Dortmund
  - Research Site, Düsseldorf
  - Research Site, Erfurt
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Göttingen
  - Research Site, Greifswald
  - Research Site, Haßloch
  - Research Site, Heidelberg
  - Research Site, Homburg
  - Research Site, Langen
  - Research Site, Leipzig
  - Research Site, Ludwigshafen
  - Research Site, Mainz
  - Research Site, Markleeberg
  - Research Site, Witten
  - Research Site, Würzburg
- Greece (8):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Chaidari, Athens
  - Research Site, Chalcis
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Thessaloniki
- Hungary (18):
  - Research Site, Balatonfüred
  - Research Site, Berettyóújfalu
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Dunaújváros
  - Research Site, Gyöngyös
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Komárom
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Sopron
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Szentes
  - Research Site, Szolnok
  - Research Site, Zalaegerszeg
- Italy (27):
  - Research Site, Ariccia
  - Research Site, Arzignano
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Cagliari
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Cona FE
  - Research Site, Cuneo
  - Research Site, Foggia
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Monza (MB)
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Piacenza
  - Research Site, Rimini
  - Research Site, Roma
  - Research Site, Rozzano MI
  - Research Site, Seriate
  - Research Site, Siena
  - Research Site, Torrette Di Ancona
  - Research Site, Trieste
  - Research Site, Vimercate MB
- Japan (74):
  - Research Site, Ichinomiya-shi, Aichi-ken
  - Research Site, Nagakute-shi, Aichi-ken
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Seto-shi, Aichi-ken
  - Research Site, Asahi-shi, Chiba
  - Research Site, Chiba, Chiba
  - Research Site, Funabashi-shi, Chiba
  - Research Site, Urayasu-shi, Chiba
  - Research Site, Imabari, Ehime
  - Research Site, Matsuyama, Ehime
  - Research Site, Chikushino-shi, Fukuoka
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kasuya-gun, Fukuoka
  - Research Site, Kitakyushu-shi, Fukuoka
  - Research Site, Koga-shi, Fukuoka
  - Research Site, Kurume-shi, Fukuoka
  - Research Site, Onga-gun, Fukuoka
  - Research Site, Fukushima, Fukushima
  - Research Site, Ogaki-shi, Gifu
  - Research Site, Maebashi, Gunma
  - Research Site, Takasaki-shi, Gunma
  - Research Site, Fukuyama-shi, Hiroshima
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Kure-shi, Hiroshima
  - Research Site, Hakodate-shi, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Amagasaki-shi, Hyōgo
  - Research Site, Himeji-shi, Hyōgo
  - Research Site, Kawanishi-shi, Hyōgo
  - Research Site, Nishinomiya-shi, Hyōgo
  - Research Site, Takarazuka-shi, Hyōgo
  - Research Site, Higashiibaraki-gun, Ibaraki
  - Research Site, Kahoku-gun, Ishikawa-ken
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Morioka, Iwate
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Hayama, Kanagawa
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Odawara-shi, Kanagawa
  - Research Site, Sagamihara-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Nankoku-shi, Kochi
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Sendai, Miyagi
  - Research Site, Nagano, Nagano
  - Research Site, Kashihara-shi, Nara
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Okayama, Okayama-ken
  - Research Site, Naha, Okinawa
  - Research Site, Shimajiri-gun, Okinawa
  - Research Site, Urasoe-shi, Okinawa
  - Research Site, Higashiosaka-shi, Osaka
  - Research Site, Matsubara-shi, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Suita-shi, Osaka
  - Research Site, Saga, Saga-ken
  - Research Site, Ureshino-shi, Saga-ken
  - Research Site, Ageo-shi, Saitama
  - Research Site, Koshigaya-shi, Saitama
  - Research Site, Wako-shi, Saitama
  - Research Site, Kusatsu-shi, Shiga
  - Research Site, Sunto-gun, Shizuoka
  - Research Site, Akishima-shi, Tokyo
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Fussa-shi, Tokyo
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Itabashi-ku, Tokyo
  - Research Site, Kodaira-shi, Tokyo
  - Research Site, Meguro-ku, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Shinjuku-ku, Tokyo
  - Research Site, Toyama, Toyama
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Vilnius
- Mexico (11):
  - Research Site, Torreón, Coahuila
  - Research Site, Pachuca, Hidalgo
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
  - Research Site, Querétaro City, Querétaro
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Culiacán, Sinaloa
  - Research Site, Xalapa, Veracruz
  - Research Site, Aguascalientes
- Netherlands (17):
  - Research Site, 's-Hertogenbosch
  - Research Site, Almelo
  - Research Site, Arnhem
  - Research Site, Breda
  - Research Site, Capelle aan den IJssel
  - Research Site, Den Helder
  - Research Site, Deventer
  - Research Site, Doetinchem
  - Research Site, Emmen
  - Research Site, Goes
  - Research Site, Groningen
  - Research Site, Leiderdorp
  - Research Site, Nijmegen
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Uden
  - Research Site, Zwolle
- New Zealand (3):
  - Research Site, Christchurch
  - Research Site, Papatoetoe, Auckland
  - Research Site, Takapuna, Auckland
- Poland (25):
  - Research Site, Bialystok
  - Research Site, Bytom
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Giżycko
  - Research Site, Kazimierza Wielka
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Kłodzko
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Miechów
  - Research Site, Oława
  - Research Site, Piotrkow Trybunalski
  - Research Site, Poznan
  - Research Site, Ruda Śląska
  - Research Site, Skierniewice
  - Research Site, Stalowa Wola
  - Research Site, Świdnik
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Włocławek
  - Research Site, Zabrze
- Portugal (6):
  - Research Site, Aveiro
  - Research Site, Coimbra
  - Research Site, Covilha
  - Research Site, Guimarães
  - Research Site, Lisbon
  - Research Site, Setúbal
- Research Site, San Juan, Puerto Rico
- Romania (9):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Piteşti
  - Research Site, Târgovişte
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Russia (20):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Ivanovo
  - Research Site, Izhevsk
  - Research Site, Kemerovo
  - Research Site, Kirov
  - Research Site, Korolyov
  - Research Site, Krasnodar
  - Research Site, Lomonosov
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Tomsk
  - Research Site, Village Novoseltsy
  - Research Site, Vladimir
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Slovakia (12):
  - Research Site, Banská Bystrica
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Rimavská Sobota
  - Research Site, Snina
  - Research Site, Svidník
  - Research Site, Trnava
- South Africa (9):
  - Research Site, Bloemfontein, Free State
  - Research Site, Parktown, Gauteng
  - Research Site, Soweto, Gauteng
  - Research Site, Sunninghill, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Umhlanga, KwaZulu-Natal
  - Research Site, Parow, Western Cape
  - Research Site, Somerset West, Western Cape
  - Research Site, Worcester, Western Cape
- Spain (19):
  - Research Site, Córdoba, Andalusia
  - Research Site, Granada, Andalusia
  - Research Site, Málaga, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Úbeda, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, San Cristóbal de La Laguna, Canary Islands
  - Research Site, Santander, Cantabria
  - Research Site, Valladolid, Castille and León
  - Research Site, Barcelona, Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Vigo, Galicia
  - Research Site, Majadahonda, Madrid
  - Research Site, El Palmar, Murcia
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Alicante, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Sweden (7):
  - Research Site, Falun
  - Research Site, Jönköping
  - Research Site, Lidköping
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Örebro
  - Research Site, Skellefteå
- Switzerland (7):
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Fribourg
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Lugano
  - Research Site, Zurich
- Turkey (Türkiye) (14):
  - Research Site, Adana
  - Research Site, Afyonkarahisar
  - Research Site, Ankara
  - Research Site, Çorum
  - Research Site, Eskişehir
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
  - Research Site, Konya
  - Research Site, Kırıkkale
  - Research Site, Mersin
  - Research Site, Sakarya
  - Research Site, Sivas
  - Research Site, Van
- Ukraine (9):
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
  - Research Site, Zaporizhzhya
- United Kingdom (32):
  - Research Site, Ayr
  - Research Site, Basingstoke
  - Research Site, Belfast
  - Research Site, Blackpool
  - Research Site, Corby
  - Research Site, Cottingham
  - Research Site, Dudley
  - Research Site, Dundee
  - Research Site, Exeter
  - Research Site, Gillingham
  - Research Site, Glasgow
  - Research Site, Harlow
  - Research Site, High Wycombe
  - Research Site, London
  - Research Site, Merthyr Tydfil
  - Research Site, Newport
  - Research Site, Northampton
  - Research Site, Northwood
  - Research Site, Norwich
  - Research Site, Peterborough
  - Research Site, Portsmouth
  - Research Site, Romford
  - Research Site, Sheffield
  - Research Site, Shipley
  - Research Site, Sidcup
  - Research Site, Solihull
  - Research Site, Stevenage
  - Research Site, Sunderland
  - Research Site, Swindon
  - Research Site, Taunton
  - Research Site, Torquay
  - Research Site, Worcester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Teerlink JR, Diaz R, Felker GM, McMurray JJV, Metra M, Solomon SD, Biering-Sorensen T, Bohm M, Bonderman D, Fang JC, Lanfear DE, Lund M, Momomura SI, O'Meara E, Ponikowski P, Spinar J, Flores-Arredondo JH, Claggett BL, Heitner SB, Kupfer S, Abbasi SA, Malik FI; GALACTIC-HF Investigators. Effect of Ejection Fraction on Clinical Outcomes in Patients Treated With Omecamtiv Mecarbil in GALACTIC-HF. J Am Coll Cardiol. 2021 Jul 13;78(2):97-108. doi: 10.1016/j.jacc.2021.04.065. Epub 2021 May 17. PMID 34015475
- [Derived] Ono R, Chimura M, Docherty KF, Jhund PS, Yang M, Henderson AD, Metra M, Liu G, Divanji PH, Heitner SB, Kupfer S, Malik FI, Felker GM, Solomon SD, Teerlink JR, McMurray JJV. Lactate Dehydrogenase and Outcomes in Patients With HF and Reduced Ejection Fraction: Insights From GALACTIC-HF. JACC Heart Fail. 2026 Jan 10:102900. doi: 10.1016/j.jchf.2025.102900. Online ahead of print. PMID 41528277
- [Derived] Lu H, Claggett BL, Felker GM, McMurray JJV, Teerlink JR, Inciardi RM, Metra M, Heitner SB, Diaz R, Malik F, Vaduganathan M, Solomon SD. Efficacy and Safety of Omecamtiv Mecarbil in Heart Failure With Reduced Ejection Fraction According to Age: The GALACTIC-HF Trial. JACC Heart Fail. 2025 Oct 22:102703. doi: 10.1016/j.jchf.2025.102703. Online ahead of print. PMID 41123512
- [Derived] Felker GM, Solomon SD, Metra M, Mcmurray JJV, Diaz R, Claggett B, Lanfear DE, Vandekerckhove H, Biering-Sorensen T, Lopes RD, Arias-Mendoza A, Momomura SI, Corbalan R, Ramires FJA, Zannad F, Heitner SB, Divanji PH, Kupfer S, Malik FI, Teerlink JR. Cardiac Troponin and Treatment Effects of Omecamtiv Mecarbil: Results From the GALACTIC-HF Study. J Card Fail. 2024 Jun;30(6):755-763. doi: 10.1016/j.cardfail.2023.11.021. Epub 2024 Jan 11. PMID 38215932
- [Derived] Pabon M, Cunningham J, Claggett B, Felker GM, McMurray JJV, Metra M, Diaz R, Wang X, Arias-Mendoza A, Bonderman D, Crespo-Leiro M, Fonseca C, Goncalvesova E, Lund M, O'Meara E, Sliwa-Hahnle K, Malik FI, Solomon SD, Teerlink JR; GALACTIC-HF Investigators. Sex Differences in Heart Failure With Reduced Ejection Fraction in the GALACTIC-HF Trial. JACC Heart Fail. 2023 Dec;11(12):1729-1738. doi: 10.1016/j.jchf.2023.07.029. Epub 2023 Oct 11. PMID 37831045
- [Derived] Docherty KF, McMurray JJV, Claggett BL, Miao ZM, Adams KF, Arias-Mendoza A, Cleland JGF, Diaz R, Echeverria Correa LE, Felker GM, Fonseca C, Li J, Metra M, Sliwa-Hahnle K, Solomon SD, Vandekerckhove HJ, Vinereanu D, Voors AA, Heitner SB, Kupfer S, Malik FI, Meng L, Teerlink JR. Efficacy of omecamtiv mecarbil in heart failure with reduced ejection fraction according to N-terminal pro-B-type natriuretic peptide level: insights from the GALACTIC-HF trial. Eur J Heart Fail. 2023 Feb;25(2):248-259. doi: 10.1002/ejhf.2763. Epub 2023 Jan 16. PMID 36597719
- [Derived] Solomon SD, Claggett BL, Miao ZM, Diaz R, Felker GM, McMurray JJV, Metra M, Corbalan R, Filippatos G, Goudev AR, Mareev V, Serpytis P, Suter T, Yilmaz MB, Zannad F, Kupfer S, Heitner SB, Malik FI, Teerlink JR. Influence of atrial fibrillation on efficacy and safety of omecamtiv mecarbil in heart failure: the GALACTIC-HF trial. Eur Heart J. 2022 Jun 14;43(23):2212-2220. doi: 10.1093/eurheartj/ehac144. PMID 35325102
- [Derived] Felker GM, Solomon SD, Claggett B, Diaz R, McMurray JJV, Metra M, Anand I, Crespo-Leiro MG, Dahlstrom U, Goncalvesova E, Howlett JG, MacDonald P, Parkhomenko A, Tomcsanyi J, Abbasi SA, Heitner SB, Hucko T, Kupfer S, Malik FI, Teerlink JR. Assessment of Omecamtiv Mecarbil for the Treatment of Patients With Severe Heart Failure: A Post Hoc Analysis of Data From the GALACTIC-HF Randomized Clinical Trial. JAMA Cardiol. 2022 Jan 1;7(1):26-34. doi: 10.1001/jamacardio.2021.4027. PMID 34643642
- [Derived] Teerlink JR, Diaz R, Felker GM, McMurray JJV, Metra M, Solomon SD, Adams KF, Anand I, Arias-Mendoza A, Biering-Sorensen T, Bohm M, Bonderman D, Cleland JGF, Corbalan R, Crespo-Leiro MG, Dahlstrom U, Echeverria LE, Fang JC, Filippatos G, Fonseca C, Goncalvesova E, Goudev AR, Howlett JG, Lanfear DE, Li J, Lund M, Macdonald P, Mareev V, Momomura SI, O'Meara E, Parkhomenko A, Ponikowski P, Ramires FJA, Serpytis P, Sliwa K, Spinar J, Suter TM, Tomcsanyi J, Vandekerckhove H, Vinereanu D, Voors AA, Yilmaz MB, Zannad F, Sharpsten L, Legg JC, Varin C, Honarpour N, Abbasi SA, Malik FI, Kurtz CE; GALACTIC-HF Investigators. Cardiac Myosin Activation with Omecamtiv Mecarbil in Systolic Heart Failure. N Engl J Med. 2021 Jan 14;384(2):105-116. doi: 10.1056/NEJMoa2025797. Epub 2020 Nov 13. PMID 33185990
- [Derived] Teerlink JR, Diaz R, Felker GM, McMurray JJV, Metra M, Solomon SD, Legg JC, Buchele G, Varin C, Kurtz CE, Malik FI, Honarpour N. Omecamtiv Mecarbil in Chronic Heart Failure With Reduced Ejection Fraction: Rationale and Design of GALACTIC-HF. JACC Heart Fail. 2020 Apr;8(4):329-340. doi: 10.1016/j.jchf.2019.12.001. Epub 2020 Feb 6. PMID 32035892
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 11,121 patients underwent screening at 944 sites in 35 countries. Of these patients, 8,256 were randomized, but 24 patients from one site were excluded because of Good Clinical Practice violations and are not included in the data reported below.
Pre-assignment Details: Participants were randomly assigned in a 1:1 ratio to receive either oral omecamtiv mecarbil (OM) or placebo.
  Randomization was stratified by randomization setting (currently hospitalized for heart failure [HF] or recently and not currently hospitalized for HF) and region (United States and Canada; Latin America; Western Europe, South Africa, and Australasia; Eastern Europe including Russia; Asia).
Groups:
- Placebo: Participants received matching placebo tablets twice a day (BID).
- Omecamtiv Mecarbil: Participants received oral omecamtiv mecarbil BID. The starting dose was 25 mg; the dose may have been adjusted at week 4 to 37.5 or 50 mg based on the predose plasma concentration measured at week 2.
Period: Overall Study
Arm/Group | Placebo | Omecamtiv Mecarbil
Started | 4112 | 4120
Received Treatment | 4101 | 4110
Completed | 3008 (7 participants in this group who discontinued the study had unknown vital status at the end of study) | 3028 (9 participants in this group who discontinued the study had unknown vital status at the end of study)
Not Completed | 1104 | 1092
Not completed — Withdrawal by Subject | 24 | 21
Not completed — Lost to Follow-up | 26 | 20
Not completed — Death | 1054 | 1051

BASELINE CHARACTERISTICS:
Population: The full analysis set included all the randomized participants except for 24 patients from a single site who were excluded on the basis of Good Clinical Practice violations.
Groups:
- Placebo: Participants received matching placebo tablets (BID).
- Total: Total of all reporting groups
Arm/Group | Placebo | Omecamtiv Mecarbil | Total
Number analyzed (Participants) | 4112 | 4120 | 8232
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (11.4) | 64.5 (11.3) | 64.5 (11.4)
Age, Customized [Count of Participants; unit: Participants]
  18 to 64 years | 1873 | 1874 | 3747
  65 to 84 years | 2211 | 2220 | 4431
  85 years and over | 28 | 26 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 874 | 875 | 1749
  Male | 3238 | 3245 | 6483
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 885 | 886 | 1771
  Not Hispanic or Latino | 3227 | 3234 | 6461
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 38 | 35 | 73
  Asian | 355 | 355 | 710
  Black or African American | 277 | 285 | 562
  Multiple | 96 | 99 | 195
  Native Hawaiian or Other Pacific Islander | 6 | 7 | 13
  White | 3201 | 3196 | 6397
  Other | 139 | 143 | 282
Randomization Setting [Count of Participants; unit: Participants]
  Currently hospitalized for heart failure | 1050 | 1051 | 2101
  Recently and not currently hospitalized for heart failure | 3062 | 3069 | 6131
Region [Count of Participants; unit: Participants]
  United States and Canada | 693 | 693 | 1386
  Latin America | 787 | 787 | 1574
  Western Europe, South Africa, and Australasia | 960 | 961 | 1921
  Eastern Europe including Russia | 1337 | 1344 | 2681
  Asia | 335 | 335 | 670

OUTCOME MEASURES:

1. Primary Outcome: Time to Cardiovascular Death or First Heart Failure Event
Description: The primary outcome was a composite of a heart-failure (HF) event or cardiovascular (CV) death, whichever occurred first, in a time-to-event analysis.
  A heart-failure event was defined as an urgent clinic visit, emergency department visit, or hospitalization for subjectively and objectively worsening heart failure leading to treatment intensification beyond a change in oral diuretic therapy.
  All deaths and HF events were adjudicated by an independent external clinical events committee (CEC) at the Duke Clinical Research Institute, using standardized definitions based on the recent American College of Cardiology/American Heart Association (ACC/AHA) standards for endpoint definitions in cardiovascular clinical trials.
  Time to cardiovascular death or first HF event was analyzed using Kaplan-Meier (KM) methods. Since the median was not calculated, the percentage of participants with a positively adjudicated event during the study is reported.
Time Frame: From randomization to up to earliest of last confirmed survival status date or analysis cut-off date (07 August 2020); the overall median duration of follow-up was 21.8 months up to a maximum of 42 months.
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Omecamtiv Mecarbil
Number analyzed (Participants) | 4112 | 4120
percentage of participants | 39.1 | 37.0
Statistical Analysis 1: Comparison: Placebo vs Omecamtiv Mecarbil; Test type: Superiority — The overall type I error was 0.05 for 2-sided testing across primary and secondary outcomes. Control for multiple comparisons was achieved using the following testing algorithm: if the primary outcome met the P-value threshold of 0.05, the alpha error would be divided unequally between cardiovascular death (96% of the overall alpha error, or 0.048) and change from baseline to week 24 in the Kansas City Cardiomyopathy Questionnaire total symptom score (4% of the overall alpha error, or 0.002); p = 0.0252, Regression, Cox; Stratified by randomization setting and region, including terms for baseline estimated glomerular filtration rate (eGFR) and treatment group; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.86 to 0.99] — Cox proportional-hazards model with baseline hazards stratified according to the randomization setting and geographic region and with the treatment group and baseline eGFR as covariates
Statistical Analysis 2: Comparison: Placebo vs Omecamtiv Mecarbil; Test type: Superiority; p = 0.0211, Stratified log-rank test; Log-rank test stratified by randomization setting and region
Statistical Analysis 3: Comparison: Placebo vs Omecamtiv Mecarbil; Competing risk subdistribution hazard ratio and associated 95% confidence intervals for treatment were computed. Deaths not included in the endpoint were considered as the competing risk; Test type: Superiority; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.86 to 0.99] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Time to Cardiovascular Death
Description: Cardiovascular death includes acute myocardial infarction (MI), sudden cardiac death, death due to heart failure, death due to stroke, death due to cardiovascular (CV) procedures, death due to CV hemorrhage, and death due to other CV causes.
  All deaths were adjudicated by an independent external clinical-events committee at the Duke Clinical Research Institute, using standardized definitions based on the recent ACC/AHA standards for endpoint definitions in cardiovascular clinical trials.
  Time to cardiovascular death was analyzed using Kaplan-Meier methods. Since the median was not calculated, the percentage of participants with a positively adjudicated event during the study is reported.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Omecamtiv Mecarbil
Number analyzed (Participants) | 4112 | 4120
percentage of participants | 19.4 | 19.6
Statistical Analysis 1: Comparison: Placebo vs Omecamtiv Mecarbil; Test type: Superiority; p = 0.8555, Regression, Cox — If significance for the primary outcome was determined, cardiovascular death was tested against an alpha of 0.048; Stratified by randomization setting and region, including terms for baseline eGFR and treatment group; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.92 to 1.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Omecamtiv Mecarbil; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.92 to 1.11] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire Total Symptom Score (KCCQ TSS) at Week 24
Description: The Kansas City Cardiomyopathy Questionnaire is a self-administered questionnaire with a 2-week recall period that includes 23 items that map to 7 domains: symptom frequency; symptom burden; symptom stability; physical limitations; social limitations; quality of life; and self-efficacy (the patient's understanding of how to manage their heart failure). The symptom frequency and symptom burden domains are merged into a total symptom score. Scores are represented on a 0-to-100-point scale, where lower scores represent more frequent and severe symptoms and scores of 100 indicate no symptoms.
  The change from baseline in KCCQ TSS was analyzed separately for each randomization setting (inpatient and outpatient).
  Least squares means are from the mixed model which includes baseline total symptom score value, region, baseline eGFR, scheduled visit, treatment group and interaction of treatment with scheduled visit as covariates.
Time Frame: Baseline and Week 24
Population: Full analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Placebo: Oupatients: Participants who had either made an urgent visit to the emergency department or been hospitalized for heart failure within 1 year before screening received placebo tablets twice a day.
- Omecamtiv Mecarbil: Outpatients: Participants who had either made an urgent visit to the emergency department or been hospitalized for heart failure within 1 year before screening received oral omecamtiv mecarbil twice daily. The starting dose was 25 mg; the dose could be adjusted at week 4 to 37.5 or 50 mg based on the predose plasma concentration measured at week 2.
- Placebo: Inpatients: Participants who were currently hospitalized for heart failure received placebo tablets twice a day.
- Omecamtiv Mecarbil: Inpatients: Participants who were currently hospitalized for heart failure received oral omecamtiv mecarbil twice daily. The starting dose was 25 mg; the dose could be adjusted at week 4 to 37.5 or 50 mg based on the predose plasma concentration measured at week 2.
Arm/Group | Placebo: Oupatients | Omecamtiv Mecarbil: Outpatients | Placebo: Inpatients | Omecamtiv Mecarbil: Inpatients
Number analyzed (Participants) | 2704 | 2715 | 835 | 868
scores on a scale | 6.29 (0.34) | 5.83 (0.34) | 21.15 (0.71) | 23.65 (0.70)
Statistical Analysis 1: Comparison: Placebo: Oupatients vs Omecamtiv Mecarbil: Outpatients; Test type: Other; Least Squares (LS) Mean Difference = -0.46, 95% CI 2-sided [-1.40 to 0.48], Standard Error of Mean 0.48 — Treatment difference = Omecamtiv mecarbil - Placebo
Statistical Analysis 2: Comparison: Placebo: Inpatients vs Omecamtiv Mecarbil: Inpatients; Test type: Other; LS Mean Difference = 2.50, 95% CI 2-sided [0.54 to 4.46], Standard Error of Mean 1.00 — Treatment difference = Omecamtiv mecarbil - Placebo
Statistical Analysis 3: Comparison: Placebo: Oupatients vs Omecamtiv Mecarbil: Outpatients vs Placebo: Inpatients vs Omecamtiv Mecarbil: Inpatients; Test type: Superiority — If significance for the primary outcome was determined, change from baseline in the KCCQ total symptom score was tested against an alpha of 0.002; p = 0.0278, Omnibus F-test
Statistical Analysis 4: Comparison: Placebo: Oupatients vs Omecamtiv Mecarbil: Outpatients vs Placebo: Inpatients vs Omecamtiv Mecarbil: Inpatients; Test type: Other; Pooled treatment difference = 0.75, 95% CI 2-sided [-2.55 to 4.51] — Overall pooled estimate of treatment difference (Omecamtiv mecarbil - Placebo) using random effects meta-analysis approach
Statistical Analysis 5: Comparison: Placebo: Oupatients vs Omecamtiv Mecarbil: Outpatients; As a sensitivity for missing data due to death, joint longitudinal and survival models were fit using KCCQ TSS observed values with random subject slopes and intercepts for the longitudinal models with terms for baseline eGFR, region, and treatment by slope. The survival models were fit for all-cause death with baseline eGFR and treatment in the proportional hazard part of the models, KCCQ TSS modeled values as the shared parameterization, stratified by region with Weibull baseline functions; Test type: Superiority; LS Mean Difference = -0.71, 95% CI 2-sided [-1.62 to 0.20] — Treatment difference = Omecamtiv mecarbil - Placebo
Statistical Analysis 6: Comparison: Placebo: Inpatients vs Omecamtiv Mecarbil: Inpatients; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; LS mean difference = 2.31, 95% CI 2-sided [0.80 to 3.82] — Treatment difference = Omecamtiv mecarbil - Placebo

4. Secondary Outcome: Time to First Heart Failure Hospitalization
Description: A HF hospitalization is defined as an event that met all of the following criteria:
  1. The participant was admitted to the hospital with a primary diagnosis of HF;
  2. The length of stay in the hospital extended for at least 24 hours;
  3. The participant exhibited documented new or worsening symptoms due to HF on presentation;
  4. The participant had objective evidence of new or worsening HF;
  5. The participant received initiation or intensification of treatment specifically for HF, including an intravenous diuretic or vasoactive agent, mechanical or surgical intervention, or mechanical fluid removal.
  Events were adjudicated by an independent external CEC at the Duke Clinical Research Institute using standardized definitions based on the ACC/AHA standards for endpoint definitions in CV clinical trials.
  Time to first HF hospitalization was analyzed using KM methods. Since the median was not calculated, the percentage of participants with a positively adjudicated event is reported.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Omecamtiv Mecarbil
Number analyzed (Participants) | 4112 | 4120
percentage of participants | 28.7 | 27.7
Statistical Analysis 1: Comparison: Placebo vs Omecamtiv Mecarbil; Test type: Superiority; p = 0.1902, Regression, Cox — If statistical significance was achieved for both the time to CV death and change from baseline in the KCCQ TSS, time to first heart failure hospitalization was to be tested at the full alpha; Stratified by randomization setting and region, including terms for baseline eGFR and treatment group; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.87 to 1.03] — Cox proportional-hazards model with baseline hazards stratified according to the randomization setting and geographic region and with the trial group and the baseline eGFR as covariates
Statistical Analysis 2: Comparison: Placebo vs Omecamtiv Mecarbil; Competing risk subdistribution hazard ratio and associated 95% confidence intervals for treatment were computed. Deaths not included in the endpoint are considered as the competing risk; Test type: Superiority; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.88 to 1.04] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Time to All-cause Death
Description: All events were adjudicated by an independent external clinical-events committee at the Duke Clinical Research Institute, using standardized definitions based on the recent ACC/AHA standards for endpoint definitions in cardiovascular clinical trials.
  Time to all-cause death was analyzed using Kaplan-Meier methods. Since the median was not calculated, the percentage of participants with an event are reported. Events that occurred up to the earliest of last confirmed survival status date or analysis cut-off date (07 August 2020) are included.
Time Frame: From randomization up to earliest of last confirmed survival status date or analysis cut-off date (07 August 2020); the overall median duration of follow-up was 21.8 months up to a maximum of 42 months.
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Omecamtiv Mecarbil
Number analyzed (Participants) | 4112 | 4120
percentage of participants | 25.9 | 25.9
Statistical Analysis 1: Comparison: Placebo vs Omecamtiv Mecarbil; Test type: Superiority; p = 0.9633, Regression, Cox — If time to first heart failure hospitalization was statistically significant, time to all-cause death was to be tested with the same alpha as time to first heart failure hospitalization; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.92 to 1.09] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from randomization until end of study (27 August 2020); median (min, max) time on study was 21.8 (0, 42) months. Adverse events are reported from first dose of study drug until 30 days after last dose; median (min, max) treatment duration was 19.5 (0, 42) months.
Description: All-cause mortality is reported for all participants randomized in the study, excluding 24 participants due to GCP violations. All-cause mortality includes all deaths that occurred during the study including any that occurred after the efficacy analysis cut-off date.
  Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Placebo | Omecamtiv Mecarbil
All-Cause Mortality (participants affected / at risk) | 1078/4112 | 1078/4120
Serious Adverse Events (participants affected / at risk) | 2435/4101 | 2373/4110
Other Adverse Events (participants affected / at risk) | 1146/4101 | 1129/4110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4101) | Omecamtiv Mecarbil (N=4110)
Anaemia (Blood and lymphatic system disorders) | 28 | 34
Anaemia of chronic disease (Blood and lymphatic system disorders) | 2 | 0
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 2 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 3
Cold type haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 2
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Normochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Splenic infarction (Blood and lymphatic system disorders) | 2 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1
Acute coronary syndrome (Cardiac disorders) | 12 | 11
Acute left ventricular failure (Cardiac disorders) | 16 | 9
Acute myocardial infarction (Cardiac disorders) | 64 | 71
Acute right ventricular failure (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 40 | 41
Angina unstable (Cardiac disorders) | 49 | 63
Aortic valve disease (Cardiac disorders) | 1 | 0
Aortic valve disease mixed (Cardiac disorders) | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 3 | 3
Arrhythmia (Cardiac disorders) | 6 | 4
Arrhythmia supraventricular (Cardiac disorders) | 3 | 4
Arteriosclerosis coronary artery (Cardiac disorders) | 7 | 2
Atrial fibrillation (Cardiac disorders) | 113 | 94
Atrial flutter (Cardiac disorders) | 25 | 23
Atrial tachycardia (Cardiac disorders) | 9 | 9
Atrial thrombosis (Cardiac disorders) | 2 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 12 | 14
Atrioventricular block second degree (Cardiac disorders) | 0 | 3
Bradyarrhythmia (Cardiac disorders) | 5 | 1
Bradycardia (Cardiac disorders) | 3 | 8
Bundle branch block left (Cardiac disorders) | 5 | 1
Cardiac amyloidosis (Cardiac disorders) | 0 | 1
Cardiac aneurysm (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 64 | 50
Cardiac asthma (Cardiac disorders) | 1 | 2
Cardiac disorder (Cardiac disorders) | 3 | 0
Cardiac failure (Cardiac disorders) | 1045 | 988
Cardiac failure acute (Cardiac disorders) | 251 | 212
Cardiac failure chronic (Cardiac disorders) | 170 | 156
Cardiac failure congestive (Cardiac disorders) | 154 | 147
Cardiac flutter (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 2 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 14 | 9
Cardiogenic shock (Cardiac disorders) | 68 | 75
Cardiomyopathy (Cardiac disorders) | 8 | 12
Cardiopulmonary failure (Cardiac disorders) | 6 | 3
Cardiorenal syndrome (Cardiac disorders) | 10 | 14
Cardiovascular insufficiency (Cardiac disorders) | 2 | 1
Chordae tendinae rupture (Cardiac disorders) | 0 | 1
Chronic left ventricular failure (Cardiac disorders) | 8 | 6
Chronotropic incompetence (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 24 | 14
Coronary artery disease (Cardiac disorders) | 24 | 26
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 10 | 6
Extrasystoles (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 3 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 8 | 9
Left ventricular dysfunction (Cardiac disorders) | 3 | 1
Left ventricular failure (Cardiac disorders) | 4 | 4
Low cardiac output syndrome (Cardiac disorders) | 3 | 2
Mitral valve incompetence (Cardiac disorders) | 8 | 9
Myocardial fibrosis (Cardiac disorders) | 3 | 2
Myocardial infarction (Cardiac disorders) | 54 | 36
Myocardial ischaemia (Cardiac disorders) | 10 | 12
Myocarditis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 3 | 2
Paroxysmal arrhythmia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 2
Pericardial haemorrhage (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 1
Pericarditis constrictive (Cardiac disorders) | 0 | 1
Postinfarction angina (Cardiac disorders) | 0 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 1
Prosthetic cardiac valve thrombosis (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 2 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 1
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 2
Sinus node dysfunction (Cardiac disorders) | 2 | 5
Sinus tachycardia (Cardiac disorders) | 2 | 2
Supraventricular extrasystoles (Cardiac disorders) | 2 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 11 | 8
Tachyarrhythmia (Cardiac disorders) | 2 | 1
Tachycardia (Cardiac disorders) | 5 | 2
Tricuspid valve incompetence (Cardiac disorders) | 1 | 1
Trifascicular block (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 18 | 24
Ventricular extrasystoles (Cardiac disorders) | 9 | 8
Ventricular fibrillation (Cardiac disorders) | 49 | 30
Ventricular flutter (Cardiac disorders) | 1 | 2
Ventricular tachyarrhythmia (Cardiac disorders) | 7 | 7
Ventricular tachycardia (Cardiac disorders) | 129 | 106
Congenital megaureter (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 1
Myocardial bridging (Congenital, familial and genetic disorders) | 1 | 0
Non-compaction cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 3
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Basedow's disease (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 3 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 4
Hypothyroidism (Endocrine disorders) | 3 | 1
Thyroiditis (Endocrine disorders) | 0 | 1
Thyrotoxic crisis (Endocrine disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 1 | 1
Arteriosclerotic retinopathy (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 9 | 8
Cataract diabetic (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Eye inflammation (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 2
Iridodialysis (Eye disorders) | 0 | 1
Iris disorder (Eye disorders) | 0 | 1
Macular fibrosis (Eye disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0
Pterygium (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Scleromalacia (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Vitreous haematoma (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 2
Abdominal adhesions (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 3
Abdominal hernia (Gastrointestinal disorders) | 3 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 13 | 6
Abdominal pain upper (Gastrointestinal disorders) | 5 | 6
Abnormal faeces (Gastrointestinal disorders) | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 2
Anal fistula (Gastrointestinal disorders) | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 3
Chronic gastritis (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1
Colitis microscopic (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 7 | 5
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 6
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 2 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 4
Enterocolitis (Gastrointestinal disorders) | 3 | 1
Epiploic appendagitis (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 5
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 2
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 7 | 4
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 2
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 14 | 18
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 3
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 2 | 1
Haemoperitoneum (Gastrointestinal disorders) | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Hernial eventration (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 3
Ileus (Gastrointestinal disorders) | 5 | 3
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 9 | 10
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1
Intestinal angina (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 4
Intestinal obstruction (Gastrointestinal disorders) | 6 | 4
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 2
Ischaemic enteritis (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 3 | 4
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3
Lower gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 | 2
Mesenteric artery embolism (Gastrointestinal disorders) | 2 | 0
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Necrotising oesophagitis (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 1
Oesophageal motility disorder (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 9
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Pancreatolithiasis (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Rectal fissure (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 3
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 10
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 6
Asthenia (General disorders) | 7 | 5
Cardiac death (General disorders) | 4 | 2
Catheter site haemorrhage (General disorders) | 0 | 1
Chest discomfort (General disorders) | 2 | 1
Chest pain (General disorders) | 22 | 15
Complication associated with device (General disorders) | 0 | 3
Death (General disorders) | 49 | 65
Discomfort (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 2
Gait disturbance (General disorders) | 1 | 0
Gait inability (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 3
Generalised oedema (General disorders) | 2 | 1
Hypothermia (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 1 | 1
Inflammation (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 1
Infusion site extravasation (General disorders) | 0 | 1
Localised oedema (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Medical device site haematoma (General disorders) | 1 | 1
Medical device site haemorrhage (General disorders) | 1 | 0
Medical device site thrombosis (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 14 | 17
Nodule (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 27 | 33
Oedema (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 7 | 8
Pacemaker generated arrhythmia (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Performance status decreased (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Physical deconditioning (General disorders) | 0 | 1
Pneumatosis (General disorders) | 1 | 0
Pyrexia (General disorders) | 6 | 3
Sudden cardiac death (General disorders) | 37 | 27
Sudden death (General disorders) | 58 | 52
Swelling face (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 3
Ulcer haemorrhage (General disorders) | 1 | 1
Vascular stent occlusion (General disorders) | 0 | 1
Vascular stent stenosis (General disorders) | 0 | 2
Vessel puncture site haemorrhage (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 2 | 1
Alcoholic liver disease (Hepatobiliary disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 6 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 1
Cardiac cirrhosis (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 6
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 9 | 11
Cholecystitis acute (Hepatobiliary disorders) | 18 | 11
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 11 | 9
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 2
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Congestive hepatopathy (Hepatobiliary disorders) | 3 | 3
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 5
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 5
Hepatic failure (Hepatobiliary disorders) | 4 | 5
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 3
Hepatic haematoma (Hepatobiliary disorders) | 2 | 0
Hepatic ischaemia (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 3
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 3 | 3
Hepatotoxicity (Hepatobiliary disorders) | 3 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 5 | 5
Jaundice (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 8 | 3
Portal hypertension (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Primary biliary cholangitis (Hepatobiliary disorders) | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 2
Heart transplant rejection (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 2
Abscess jaw (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 4 | 2
Acute endocarditis (Infections and infestations) | 1 | 1
Acute hepatitis B (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 3 | 3
Appendiceal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 3 | 4
Appendicitis perforated (Infections and infestations) | 3 | 1
Arteriosclerotic gangrene (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 2 | 2
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 6 | 4
Bacterial infection (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 3 | 3
Bacterial tracheitis (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 3
Bronchitis (Infections and infestations) | 24 | 25
Bronchitis bacterial (Infections and infestations) | 1 | 3
Bronchitis viral (Infections and infestations) | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Burn infection (Infections and infestations) | 2 | 0
Bursitis infective staphylococcal (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 3 | 8
COVID-19 pneumonia (Infections and infestations) | 3 | 7
Catheter bacteraemia (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 24 | 34
Chagas' cardiomyopathy (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Citrobacter sepsis (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0
Clostridial sepsis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 2
Clostridium difficile infection (Infections and infestations) | 2 | 3
Complicated appendicitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 5 | 3
Device related sepsis (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 2 | 6
Diabetic gangrene (Infections and infestations) | 1 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 4
Eczema infected (Infections and infestations) | 1 | 0
Embolic pneumonia (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 7 | 3
Endocarditis bacterial (Infections and infestations) | 1 | 2
Endocarditis enterococcal (Infections and infestations) | 0 | 2
Enterobacter bacteraemia (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Enterocolitis bacterial (Infections and infestations) | 2 | 0
Enterocolitis viral (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 9 | 10
Escherichia infection (Infections and infestations) | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 2 | 0
Fournier's gangrene (Infections and infestations) | 2 | 0
Fungal infection (Infections and infestations) | 1 | 0
Gallbladder abscess (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 8 | 5
Gas gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 11 | 15
Gastroenteritis bacterial (Infections and infestations) | 1 | 2
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Graft infection (Infections and infestations) | 1 | 1
Groin abscess (Infections and infestations) | 0 | 1
Hepatitis A (Infections and infestations) | 1 | 0
Hepatitis viral (Infections and infestations) | 0 | 1
Herpes dermatitis (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Implant site infection (Infections and infestations) | 1 | 3
Incision site abscess (Infections and infestations) | 1 | 0
Infected seroma (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 5 | 2
Infection (Infections and infestations) | 6 | 2
Infectious pleural effusion (Infections and infestations) | 1 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 | 4
Infective myositis (Infections and infestations) | 0 | 1
Infective spondylitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 15 | 19
Intervertebral discitis (Infections and infestations) | 2 | 0
Jejunal gangrene (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 2
Large intestine infection (Infections and infestations) | 1 | 1
Laryngitis (Infections and infestations) | 0 | 2
Liver abscess (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 6 | 3
Lower respiratory tract infection (Infections and infestations) | 6 | 7
Lower respiratory tract infection viral (Infections and infestations) | 2 | 1
Lung abscess (Infections and infestations) | 0 | 1
Lymphadenitis bacterial (Infections and infestations) | 1 | 0
Mediastinitis (Infections and infestations) | 0 | 1
Medical device site infection (Infections and infestations) | 3 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 1
Myiasis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 12 | 8
Osteomyelitis acute (Infections and infestations) | 0 | 1
Osteomyelitis bacterial (Infections and infestations) | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 1
Otitis media bacterial (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 5 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 179 | 171
Pneumonia adenoviral (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 6 | 7
Pneumonia escherichia (Infections and infestations) | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 2 | 0
Pneumonia klebsiella (Infections and infestations) | 2 | 1
Pneumonia moraxella (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 2
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 2
Prostatic abscess (Infections and infestations) | 1 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 4 | 6
Pulmonary tuberculosis (Infections and infestations) | 4 | 2
Pyelonephritis (Infections and infestations) | 5 | 2
Pyelonephritis acute (Infections and infestations) | 4 | 3
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 24 | 15
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection fungal (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 2 | 0
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 60 | 51
Sepsis syndrome (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 32 | 37
Sinusitis (Infections and infestations) | 1 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 2
Skin graft infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 1
Soft tissue infection (Infections and infestations) | 1 | 4
Staphylococcal bacteraemia (Infections and infestations) | 2 | 3
Staphylococcal infection (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 5 | 2
Sternitis (Infections and infestations) | 1 | 0
Stitch abscess (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Streptococcal endocarditis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 4 | 3
Tuberculoma of central nervous system (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 11 | 14
Urinary tract infection (Infections and infestations) | 32 | 33
Urinary tract infection bacterial (Infections and infestations) | 6 | 3
Urinary tract infection enterococcal (Infections and infestations) | 2 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0
Urogenital infection bacterial (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 15 | 7
Vascular device infection (Infections and infestations) | 1 | 1
Viraemia (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 3 | 3
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Wound abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 5 | 1
Wound infection bacterial (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Wound sepsis (Infections and infestations) | 1 | 2
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 5 | 4
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 2
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Cardiac vein perforation (Injury, poisoning and procedural complications) | 1 | 0
Cataract traumatic (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 3
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 2
Dialysis disequilibrium syndrome (Injury, poisoning and procedural complications) | 1 | 0
Epidural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Eschar (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 10
Femoral neck fracture (Injury, poisoning and procedural complications) | 8 | 8
Femur fracture (Injury, poisoning and procedural complications) | 14 | 11
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 5 | 7
Humerus fracture (Injury, poisoning and procedural complications) | 4 | 6
Hyphaema (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 3
Injury corneal (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 3
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 2
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 3
Osteophyte fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Pneumocephalus (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 3
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 5
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 2 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 2 | 2
Rib fracture (Injury, poisoning and procedural complications) | 7 | 6
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 4
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 3
Subdural haematoma (Injury, poisoning and procedural complications) | 9 | 8
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 2 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 | 5
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 2
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 0 | 1
Vena cava injury (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 2
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 3 | 2
Anticoagulation drug level above therapeutic (Investigations) | 1 | 5
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood calcium decreased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood glucose decreased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Cardiac output decreased (Investigations) | 1 | 2
Catheterisation cardiac (Investigations) | 0 | 1
Coagulation time prolonged (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1
HIV antibody positive (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme abnormal (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 6 | 4
Influenza A virus test positive (Investigations) | 1 | 1
International normalised ratio abnormal (Investigations) | 1 | 0
International normalised ratio decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 2 | 3
Liver function test abnormal (Investigations) | 0 | 4
Liver function test increased (Investigations) | 2 | 2
Oxygen consumption increased (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 1 | 3
Staphylococcus test positive (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 3
Transplant evaluation (Investigations) | 0 | 1
Troponin increased (Investigations) | 1 | 3
Weight decreased (Investigations) | 2 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 15 | 19
Diabetes mellitus (Metabolism and nutrition disorders) | 8 | 15
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 | 6
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 | 3
Diabetic ketosis (Metabolism and nutrition disorders) | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 8 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 7 | 3
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 7 | 14
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 9
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 21 | 20
Hyperosmolar state (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 13 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 7
Hypokalaemic syndrome (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 19 | 14
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 3
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 6 | 2
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 2
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Elbow deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 10
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 12
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenosquamous cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 6
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine tumour of the lung metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Alcohol induced persisting dementia (Nervous system disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 1
Amnesia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Brain compression (Nervous system disorders) | 0 | 1
Brain hypoxia (Nervous system disorders) | 0 | 1
Brain injury (Nervous system disorders) | 2 | 2
Brain oedema (Nervous system disorders) | 0 | 2
Brain stem stroke (Nervous system disorders) | 2 | 1
Carotid arteriosclerosis (Nervous system disorders) | 1 | 1
Carotid artery disease (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 3 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 1 | 0
Cerebral circulatory failure (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 7 | 2
Cerebral hypoperfusion (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 13 | 8
Cerebral ischaemia (Nervous system disorders) | 4 | 3
Cerebrovascular accident (Nervous system disorders) | 29 | 25
Cerebrovascular disorder (Nervous system disorders) | 0 | 2
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 1
Cognitive disorder (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 0 | 1
Complex regional pain syndrome (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 8 | 6
Dizziness postural (Nervous system disorders) | 3 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 1
Embolic stroke (Nervous system disorders) | 1 | 2
Encephalopathy (Nervous system disorders) | 2 | 2
Epilepsy (Nervous system disorders) | 2 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 7 | 3
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 4 | 1
Hemianopia (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 0 | 1
Hyperglycaemic unconsciousness (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 7 | 2
Ischaemic stroke (Nervous system disorders) | 38 | 36
Lacunar infarction (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 2 | 2
Meningism (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 5 | 5
Mononeuritis (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neuromyopathy (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 2
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Orthostatic intolerance (Nervous system disorders) | 2 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Post-traumatic epilepsy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 5 | 8
Psychogenic seizure (Nervous system disorders) | 1 | 0
Psychomotor disadaptation syndrome (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Radicular pain (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 2
Seizure like phenomena (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1
Stroke in evolution (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 6 | 3
Syncope (Nervous system disorders) | 46 | 42
Thrombotic stroke (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 24 | 17
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Vertigo CNS origin (Nervous system disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Device alarm issue (Product Issues) | 0 | 1
Device dislocation (Product Issues) | 2 | 0
Device electrical impedance issue (Product Issues) | 1 | 0
Device extrusion (Product Issues) | 1 | 1
Device inappropriate shock delivery (Product Issues) | 1 | 1
Device lead damage (Product Issues) | 1 | 0
Device lead issue (Product Issues) | 1 | 0
Device leakage (Product Issues) | 1 | 0
Device malfunction (Product Issues) | 6 | 6
Device occlusion (Product Issues) | 0 | 2
Device physical property issue (Product Issues) | 1 | 0
Device power source issue (Product Issues) | 1 | 3
Device signal detection issue (Product Issues) | 0 | 1
Device stimulation issue (Product Issues) | 1 | 2
Lead dislodgement (Product Issues) | 0 | 2
Oversensing (Product Issues) | 1 | 0
Undersensing (Product Issues) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 1
Behaviour disorder (Psychiatric disorders) | 1 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Communication disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 4 | 2
Confusional state (Psychiatric disorders) | 1 | 2
Conversion disorder (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 4 | 2
Disorientation (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 2 | 0
Mental disorder (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 4 | 2
Panic attack (Psychiatric disorders) | 0 | 1
Personality disorder (Psychiatric disorders) | 1 | 0
Psychotic behaviour (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 2
Suicide attempt (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 138 | 129
Anuria (Renal and urinary disorders) | 1 | 1
Atonic urinary bladder (Renal and urinary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 36 | 36
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
End stage renal disease (Renal and urinary disorders) | 4 | 7
Haematinuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 7 | 3
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 2
Hypertensive nephropathy (Renal and urinary disorders) | 1 | 0
Micturition disorder (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 5 | 1
Nephropathy (Renal and urinary disorders) | 1 | 2
Oliguria (Renal and urinary disorders) | 0 | 1
Postrenal failure (Renal and urinary disorders) | 1 | 3
Renal arteriosclerosis (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal artery thrombosis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 31 | 25
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 29 | 25
Renal infarct (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 4
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 | 5
Epididymal cyst (Reproductive system and breast disorders) | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 2 | 0
Spermatocele (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 18 | 20
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 38 | 63
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 28
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 | 11
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13 | 20
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 12 | 14
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 18 | 22
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 6 | 4
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Peau d'orange (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 | 6
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Physical assault (Social circumstances) | 0 | 1
Victim of homicide (Social circumstances) | 1 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 1
Arrhythmia prophylaxis (Surgical and medical procedures) | 0 | 1
Bladder catheter replacement (Surgical and medical procedures) | 1 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 1
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 | 3
Coronary angioplasty (Surgical and medical procedures) | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 0 | 1
Coronary revascularisation (Surgical and medical procedures) | 2 | 2
Heart transplant (Surgical and medical procedures) | 2 | 2
Hernia diaphragmatic repair (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 2 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 2 | 0
Implantable defibrillator removal (Surgical and medical procedures) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 2 | 0
Preoperative care (Surgical and medical procedures) | 0 | 1
Toe amputation (Surgical and medical procedures) | 2 | 1
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 5 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 2
Aortic dissection (Vascular disorders) | 1 | 0
Aortic dissection rupture (Vascular disorders) | 1 | 0
Aortic rupture (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 4 | 1
Arterial disorder (Vascular disorders) | 0 | 2
Arterial haemorrhage (Vascular disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arterial perforation (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 2 | 4
Axillary vein thrombosis (Vascular disorders) | 1 | 0
Brachiocephalic vein thrombosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 7 | 0
Diabetic macroangiopathy (Vascular disorders) | 0 | 1
Distributive shock (Vascular disorders) | 1 | 0
Dry gangrene (Vascular disorders) | 0 | 1
Embolism arterial (Vascular disorders) | 0 | 3
Extremity necrosis (Vascular disorders) | 3 | 3
Haematoma (Vascular disorders) | 4 | 2
Haemodynamic instability (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 10 | 9
Hypertensive crisis (Vascular disorders) | 5 | 3
Hypertensive emergency (Vascular disorders) | 2 | 1
Hypertensive urgency (Vascular disorders) | 1 | 4
Hypoperfusion (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 37 | 49
Hypovolaemic shock (Vascular disorders) | 4 | 5
Iliac artery stenosis (Vascular disorders) | 0 | 1
Infarction (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Leriche syndrome (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 1 | 0
Orthostatic hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 11 | 12
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 18 | 17
Peripheral artery occlusion (Vascular disorders) | 5 | 2
Peripheral artery stenosis (Vascular disorders) | 2 | 2
Peripheral artery thrombosis (Vascular disorders) | 2 | 6
Peripheral ischaemia (Vascular disorders) | 14 | 9
Peripheral vascular disorder (Vascular disorders) | 3 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Post thrombotic syndrome (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Varicose vein ruptured (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 2 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4101) | Omecamtiv Mecarbil (N=4110)
Cardiac failure (Cardiac disorders) | 291 | 268
Hyperkalaemia (Metabolism and nutrition disorders) | 213 | 202
Dizziness (Nervous system disorders) | 183 | 232
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 258 | 249
Hypertension (Vascular disorders) | 222 | 190
Hypotension (Vascular disorders) | 242 | 276

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT02929329/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT02929329/SAP_001.pdf